CLINICAL TRIAL: NCT01098643
Title: Patient Satisfaction With Placement of Implantable Venous Access Devices
Brief Title: Satisfaction With Placement of Implantable Venous Access Devices in Patients With Solid Tumors
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: not enough pts for available to reach goal
Sponsor: Vanderbilt University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Kristin Ancell, MD, Vanderbilt University
Organization: Vanderbilt University Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Purpose: Health Services Research
Other Study IDs: CDR0000669012; P30CA068485 (NIH); VU-VICC-SUPP-0982
Record Dates: First submitted 2010-04-02; First posted 2010-04-05 (Estimated); Last update posted 2017-04-04 (Actual); Status verified 2010-03

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: computer-assisted intervention
Other: medical chart review
Other: questionnaire administration
Other: survey administration

SUMMARY:
RATIONALE: Gathering information about patients with solid tumors who have implantable venous access devices may help doctors learn more about patient satisfaction.

PURPOSE: This phase I trial is studying satisfaction with placement of implantable venous access devices in patients with solid tumors.

DETAILED DESCRIPTION:
OBJECTIVES:

* To determine patient satisfaction with subcutaneous venous-access device placement in oncology patients.

OUTLINE: Patients complete a computer-based survey while in the treatment area of the Vanderbilt Oncology Clinic. Basic demographic information and basic information regarding the placement of the device and complications are collected from the patient's medical record.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of a solid tumor malignancy

  * No hematological malignancy
* Patient at the Vanderbilt Oncology Clinic
* Has undergone placement of a subcutaneous, single-lumen venous-access device within the past 6 months

  * No patients who have had ≥ 2 venous-access devices placed by ≥ 1 department

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* Not currently undergoing preparation for or process of stem cell transplantation

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2009-10 (Actual); Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Overall satisfaction with port placement | n/a - study closed

SECONDARY OUTCOMES:
Frequency of complications
Frequency of port failure
Need for removal of device

CONTACTS AND LOCATIONS:
Overall Officials: Kristin Ancell, MD, Principal Investigator — Vanderbilt-Ingram Cancer Center
Locations (2):
- United States (2):
  - Vanderbilt-Ingram Cancer Center - Cool Springs, Nashville, Tennessee
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: No
never published, terminated